CLINICAL TRIAL: NCT02826837
Title: A Phase I/IIa Dose-Escalation Study Evaluating the Safety, Tolerability and Efficacy of LEAC-102 in Combination With FOLFOX + Bevacizumab/Cetuximab in Subjects With Advanced Colorectal Cancer
Brief Title: LEAC-102 for Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taiwan Leader Biotech Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEAC-102-01
Record Dates: First submitted 2016-06-07; First posted 2016-07-11 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: Advanced Colorectal Cancer
MeSH Terms: interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEAC-102 and FOLFOX+Bevacizumab/Cetuximab (Experimental): The subjects will be administered folinic acid (Leucovorin; LV), Fluorouracil (5-FU) and Oxaliplatin (FOLFOX) + Bevacizumab/Cetuximab by intravenous infusion.
  Cycles repeat every 2 weeks. Dose and schedule modifications may be made at the treating physician's discretion.
  A standard 3+3 trial design will be used for LEAC-102 dose escalation cohorts.The dosing of LEAC-102 will be divided into 3 cohorts, the subjects will receive LEAC-102 every day
  Cohort 1: LEAC-102 500 mg capsule, 3 capsules, three times per day for 24 weeks (oral), Cohort 2: LEAC-102 500 mg capsule, 4 capsules, three times per day for 24 weeks (oral), Cohort 3: LEAC-102 500 mg capsule, 5 capsules, three times per day for 24 weeks (oral)
  Interventions: Drug: LEAC-102 500mg capsule and FOLFOX + Bevacizumab/Cetuximab

INTERVENTIONS:
Drug: LEAC-102 500mg capsule and FOLFOX + Bevacizumab/Cetuximab — The subjects will be administered FOLFOX + Bevacizumab/Cetuximab by intravenous infusion.
  Cycles repeat every 2 weeks. Dose and schedule modifications may be made at the treating physician's discretion.
  A standard 3+3 trial design will be used for LEAC-102 dose escalation cohorts.The dosing of LEAC-102 will be divided into 3 cohorts, the subjects will receive LEAC-102 every day
  Cohort 1: LEAC-102 500 mg capsule, 3 capsules, three times per day for 24 weeks (oral), Cohort 2: LEAC-102 500 mg capsule, 4 capsules, three times per day for 24 weeks (oral), Cohort 3: LEAC-102 500 mg capsule, 5 capsules, three times per day for 24 weeks (oral)

SUMMARY:
A Phase I/IIa Dose-Escalation Study Evaluating the Safety, Tolerability and Efficacy of LEAC-102 in Combination with FOLFOX + Bevacizumab/Cetuximab in Subjects with Advanced Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged at least 20 years old
2. Histologically or cytologically confirmed measurable and/or evaluable advanced (stage III/IV) colorectal cancer that can be accurately assessed by CT/MRI scan (RECIST v1.1) for which regimen of FOLFOX + Bevacizumab/Cetuximab is arranged by the investigator
3. Subjects may be treatment naïve, or may have received therapy for colorectal cancer.
4. ECOG performance status ≤ 2 and life expectancy ≥ 12 months Note: ECOG = Eastern Cooperative Oncology Group
5. Dated and signed informed consent

Exclusion Criteria:

1. Primary CNS malignancies or clinically active CNS metastases Note: CNS = central nervous system
2. Ascertained hypersensitivity to any component of investigational product or FOLFOX + Bevacizumab/Cetuximab that the subject will be treated
3. Any of the following hematologic abnormalities:

   1. Hemoglobin < 10.0 g/dL,
   2. ANC < 1,500/μL,
   3. Platelets < 100,000 /μL Note: ANC = absolute neutrophil count
4. Any of the following serum chemistry abnormalities:

   1. Total bilirubin > 1.5 × ULN,
   2. AST or ALT > 2.5 × ULN,
   3. Gamma-GT > 2.5 x ULN,
   4. Alk-P > 2.5 x ULN,
   5. serum albumin < 3.0 g/dL,
   6. creatinine > 1.5 × ULN,
   7. any other ≥ Grade 3 laboratory abnormality at baseline (other than those listed above)

   Note: ULN = upper limit of normal. AST = aspartate transaminase, ALT: alanine transaminase, Gamma-GT = Gamma-glutamyl transferase, Alk-P = alkaline phosphatase
5. Requirement for ongoing systemic steroid, or immunosuppressive agents
6. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral LEAC-102 treatment
7. Active clinically serious infection
8. Known history of HIV or hepatitis B or C Note: HIV = human immunodeficiency virus
9. Uncontrolled psychiatric disorder or altered mental status precluding informed consent or necessary testing
10. Consumption of herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) within 2 weeks prior to the start of Cycle 1 of FOLFOX + Bevacizumab/Cetuximab administration
11. Significant cardiovascular disease, including:

    1. Active clinically symptomatic left ventricular failure
    2. Active hypertension (diastolic blood pressure > 100 mmHg). Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 4 weeks prior to start of Cycle 1 of FOLFOX + Bevacizumab/Cetuximab administration
    3. Uncontrolled hypertension: Blood pressure >140/90 mmHg on more than 2 antihypertensive medications
    4. Myocardial infarction, severe angina, or unstable angina within 12 weeks prior to start of Cycle 1 of FOLFOX + Bevacizumab/Cetuximab administration
    5. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
12. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent
13. Has received an investigational agent within 4 weeks of entering this study
14. With any condition judged by the investigator that entering the trial may be detrimental to the subject

15 Female with childbearing potential who is lactating or has positive urine pregnancy test at Screening visit

16. Subject with either gender refuses to adopt at least two forms of birth control (at least one of which must be a barrier method) during the study and until 30 days after study treatment.

Note: Acceptable forms include:

1. Established use of oral, injected or implanted hormonal methods of contraception.
2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
3. Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

17. Subjects with grade 2 or above chronic neuropathy

18. Subjects with known dihydropyrimidine dehydrogenase (DPD) deficiency.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Week 4
  First two cycles of FOLFOX + Bevacizumab/Cetuximab for advanced Colorectal Cancer (cycle length = 2 weeks)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Incidence of serious adverse events (SAEs) | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Response rate | Week 24
Progression free survival | Week 24
Overall survival | Week 24
Incidences of myelosuppression | Weeks Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Change in white blood cells (WBCs) level at all post-treatment visits compared to baseline | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Change in platelet level at all post-treatment visits compared to baseline | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Change in hemoglobin level at all post-treatment visits compared to baseline | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Change in serum inflammatory cytokines level at all post-treatment visits compared to baseline | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Change in serum c-reactive protein level at all post-treatment visits compared to baseline | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24
Changes in global health/QoL standardized score at post-treatment visits compared to baseline | Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22,24